CLINICAL TRIAL: NCT06354530
Title: Neoadjuvant Immunotherapy Plus Chemotherapy and Anlotinib Versus Immunotherapy Combined With Concurrent Chemoradiotherapy in the Treatment of Locally Advanced ESCC
Brief Title: A Study of Neoadjuvant Therapy for the Treatment of Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Army Medical Center of PLA (Other Government)
Responsible Party: Principal Investigator, Mengxia Li, Department of Cancer Center, Army Medical Center of PLA, Army Medical Center of PLA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023 (315)
Record Dates: First submitted 2024-03-18; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Neoadjuvant Therapy; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — anlotinib; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant immunotherapy plus chemotherapy and anlotinib (Experimental): neoadjuvant immunotherapy plus chemotherapy and anlotinib
  Interventions: Radiation: Thoracic radiotherapy
- neoadjuvant immunotherapy combined with concurrent chemoradiotherapy (Experimental): neoadjuvant immunotherapy combined with concurrent chemoradiotherapy
  Interventions: Drug: anlotinib

INTERVENTIONS:
Drug: anlotinib — Drug: Camrelizumab 200mg on Day 1 of each 3-week cycle for 2 cycles during the neoadjuvant period
  Drug: Carboplatin Area under the curve of 5 on Day 1 of each 3-week cycle for 2 cycles
  Drug: Cisplatin 75 mg/m2 on Day 1 of each 3-week cycle, for 2 cycles
  Drug: Paclitaxel 135-175 mg/m2 on Day 1 of each 3-week cycle for 2 cycles
  Drug: Nab-Paclitaxel 220-260 mg/m2 on Day 1 of each 3-week cycle for 2 cycles
  Drug: anlotinib 8 mg/day orally (from days 1 to 14 in a 21-day cycle) for 2 cycles
  Arms: neoadjuvant immunotherapy combined with concurrent chemoradiotherapy
Radiation: Thoracic radiotherapy — Drug: Camrelizumab 200mg on Day 1 of each 3-week cycle for 2 cycles during the neoadjuvant period
  Drug: Carboplatin Area under the curve of 5 on Day 1 of each 3-week cycle for 2 cycles
  Drug: Cisplatin 75 mg/m2 on Day 1 of each 3-week cycle, for 2 cycles
  Drug: Paclitaxel 135-175 mg/m2 on Day 1 of each 3-week cycle for 2 cycles
  Drug: Nab-Paclitaxel 220-260 mg/m2 on Day 1 of each 3-week cycle for 2 cycles
  Thoracic radiotherapy RT once daily (from cycle 1 [C1D1], 41.4Gy/23Fx, 1.8Gy daily, for 4.6 weeks, 5 days/week)
  Other Names: radiotherapy
  Arms: neoadjuvant immunotherapy plus chemotherapy and anlotinib

SUMMARY:
The goal of this interventional study is to compare the safety and efficacy of neoadjuvant immunotherapy plus chemotherapy and anlotinib versus immunotherapy combined with concurrent chemoradiotherapy in the treatment of locally advanced esophageal squamous cell carcinoma. The main question it aims to answer is: To evaluate the safety and efficacy of neoadjuvant immunotherapy plus chemotherapy and anlotinib versus immunotherapy combined with concurrent chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma and to explore the optimal preoperative neoadjuvant treatment regimen for esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
The goal of this single-center, open-label, non-inferior, randomized controlled, interventional study is to compare the safety and efficacy of neoadjuvant immunotherapy plus chemotherapy and anlotinib versus immunotherapy combined with concurrent chemoradiotherapy in the treatment of locally advanced esophageal squamous cell carcinoma. The main question it aims to answer is: To evaluate the safety and efficacy of neoadjuvant immunotherapy plus chemotherapy and anlotinib versus immunotherapy combined with concurrent chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma and to explore the optimal preoperative neoadjuvant treatment regimen for esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Surgically resectable cT1-4aN+M0 or cT3-4aN0M0 esophageal squamous cell carcinoma initially diagnosed by histology or cytology
* Patients who can take anlotinib capsules orally
* No previous systematic antitumor treatment
* ECOG PS 0-1
* The function of important organs meets the following requirements: absolute neutrophil count≥1.5×10^9 / L; platelet≥80×10^9 / L; hemoglobin≥80×10^9 / L; total bilirubin≤1.5×upper limit of normal; within normal serum creatinine; ALT and glutamatergic aminase≤2.5× upper limit of normal
* No incurable serious complications or other major diseases
* The thoracic surgeon judges that the operation can be tolerated
* Female subjects with fertility, and male subjects with childbearing partners, required a medically approved contraceptive during study treatment and at least 6 months after the last chemotherapy
* The subjects volunteered to join the study, signed informed consent, had good compliance and cooperated with follow-up

Exclusion Criteria:

* BMI<18.5kg/m2 or 10% weight loss in 2 months before screening (while considering the effect of large chest ascites on body weight)
* Patients with tracheal / bronchial / macrovascular invasion, deep ulcer esophagus, digestive tract perforation and / or fistula, major bleeding, and poor lung function or previous chronic lung disease within 6 months prior to initial medication
* Patients with significant feeding obstruction unable to take oral anlotinib
* Known history of allergy to any component of biological or PD-1 mab formulation, albumin-bound paclitaxel, carboplatin and other platinum drugs manufactured by Chinese hamster ovary cells (CHO)
* Have received any of the following treatments: any investigational drug; enrolled in another clinical study except for an observational (non-interventional) clinical study; received anti-tumor or live vaccine
* A history of active autoimmune diseases and autoimmune diseases
* A history of immunodeficiency, including a positive HIV test, or other acquired, congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation
* The subject had cardiovascular clinical symptoms or disease that were not well controlled
* Patients with active hepatitis B or hepatitis C and active pulmonary tuberculosis
* Severe infection (CTCAE> 2) occurred within 4 weeks prior to initial use of study drug, such as severe pneumonia, bacteremia, infection requiring hospitalization; baseline chest imaging indicated active lung inflammation, symptoms and signs of infection within 2 weeks prior to initial use of study drug or the need for oral or intravenous antibiotics, except for prophylactic antibiotics
* Major surgery (except diagnostic surgery) within 28 days prior to treatment, or is expected to undergo major surgery during the study
* Any other malignancy had been diagnosed within 5 years prior to the first use of study drug, except for nausea tumors with low risk and mortality (5-year survival> 90%), such as adequately treated basal or squamous cell skin carcinoma or carcinoma of the cervix
* Female patients during pregnancy or lactation and who were refused or unable to use contraception
* At the discretion of the investigator, the subject had other factors that could contribute to his forced termination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR), Major pathological response (MPR) | Up to approximately 15 weeks after randomization
  Defined as the lack of any viable tumour cells after complete evaluation in the resected lung cancer specimen and all sampled regional lymph nodes
Major pathological response (MPR) | Up to approximately 15 weeks after randomization
  Major pathological response (MPR)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 15 weeks after randomization
  Objective response rate (ORR)
3-year disease free survival | From date of randomization to approximately 3 years after date of resection
  3-year disease free survival
R0 excision rate | Up to approximately 15 weeks after randomization
  R0 excision rate
3-year overall survival | From date of randomization to approximately 3 years after date of resection
  3-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing Wang, Principal Investigator — Army Medical Center of PLA
Locations (1):
- Army Medical Center of PLA, Chongqing, None Selected, China